CLINICAL TRIAL: NCT02790450
Title: Acute Effects of Benzbromaron on the Pulmonary Circulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27-253 ex 14/15
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Benzbromarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Benzbromarone (Experimental): 1x200mg Benzbromarone
  Interventions: Drug: Benzbromarone

INTERVENTIONS:
Drug: Benzbromarone — 1x200mg Benzbromarone will be applied after baseline measurements during right heart catheterization. The effects of the drug on the pulmonary hemodynamics will be assessed after 2 hours.

SUMMARY:
Actual studies suggest that a calcium activated chlorid channel (TMEM16A) may play a relevant role in the pathogenesis of pulmonary arterial hypertension (PAH). The inhibition of this channel led to pulmonary vasorelaxation in preclinical studies. Benzbromarone is a well known inhibitor of the TMEM16A channel and is used in patients with gout.

In this pilot study the investigators plan to investigate if Benzbromarone has an acute effect on the pulmonary arteries in humans. This will be investigated within the frame of a right heart catheterization performed in patients with known PAH due to clinical reasons. The investigators hypothesize that the application of Benzbromarone leads to pulmonary vasodilation, which can be recognized by the decrease in pulmonary vascular resistance. In addition, the change in pulmonary and systemic arterial pressure, pulmonary arterial wedge pressure, heart rate and arterial oxygen saturation will be assessed. Due to clinical reasons patients will receive NO (15 ppm) during right heart catheterization. Hemodynamic changes upon NO and Benzbromarone may be compared.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* known pulmonary arterial hypertension
* right heart catheterization indicated due to clinical reasons

Exclusion Criteria:

* known allergy against Benzbromaron, Gelborange S or other ingredient of the used drug (Benzbromarone AL) or a drug with similar chemical structure
* severe renal insufficiency (GFR<30ml/min/kg)
* renal diathesis
* severe hepatic disease (Bilirubin >1.6 mg% or AST or ALT > 3x Norm)
* known pregnancy
* uncontrolled systemic arterial hypertension (>150 mmHg systolic or 95 mmHg diastolic)
* uncontrolled ventricular arrythmia
* uncontrolled bradycardic or tachycardic supraventricular arrythmia
* myocardiac infarction within the last 12 months
* pulmonary embolism within the last 6 months
* ongoing iv. or sc. Prostanoid therapy for PAH
* Pulmonary hypertension other than PAH

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (Wood units) assessed by right heart catheterization | 2 hours

SECONDARY OUTCOMES:
Mean pulmonary arterial pressure (mmHg) assessed by right heart catheterization | 2 hours
Mean systemic arterial pressure (mmHg) assessed by sphygmomanometer | 2 hours
arterial oxygen saturation 8%) assessed by arterial blood gas analysis | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes